CLINICAL TRIAL: NCT07337161
Title: Stereotactic Post-operative Radiotherapy for Intraparotid Metastatic Cutaneous Squamous Cell Carcinoma
Acronym: SPRINT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: David Palma (Other)
Responsible Party: Sponsor-Investigator, David Palma, Professor, Schulich School of Medicine & Dentistry, University of Western Ontario, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Organization: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5201; 15521 (Other: London Health Science Centre (LHSCRI))
Record Dates: First submitted 2025-08-28; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Cutaneous; Head and Neck Cancer Squamous Cell Carcinoma
Keywords: skin; head and neck; radiation; SBRT; SABR

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1: Control (Active Comparator): Patients in Arm 1 will receive daily conventional fractionation radiation over 4 or 6-6.5 weeks based on the treating oncologist's discretion. The below dose levels are recommended in the following clinical scenarios but may be modified per institutional standards:
  20-fraction regimen or 30 to 33-fraction regimen
  Interventions: Radiation: Standard Radiation
- Arm 2: SBRT arm (Experimental): Patients in Arm 2 will receive ultra-hypofractionated stereotactic radiation over 5 treatments delivered every other weekday or twice weekly as follows:
  * 40 to 42.5 Gy in 5 fractions: any areas of gross residual disease, or gross PNI on imaging
  * 32.5 to 35 Gy in 5 fractions: microscopic areas at risk including positive margin and/or ENE
  * 30 Gy in 5 fractions: entire operative bed including areas of primary tumor and involved nodes and dissected cervical nodal levels
  * 27.5 to 30 Gy 5 fractions: at risk undissected cervical nodal levels adjacent to pathologically involved nodal levels, based on the discretion of the treating oncologist
  Interventions: Radiation: SBRT

INTERVENTIONS:
Radiation: SBRT — Patients will receive ultra-hypofractionated stereotactic radiation over 5 treatments delivered every other weekday or twice weekly as follows:
  * 40 to 42.5 Gy in 5 fractions: any areas of gross residual disease, or gross PNI on imaging
  * 32.5 to 35 Gy in 5 fractions: microscopic areas at risk including positive margin and/or ENE
  * 30 Gy in 5 fractions: entire operative bed including areas of primary tumor and involved nodes and dissected cervical nodal levels
  * 27.5 to 30 Gy 5 fractions: at risk undissected cervical nodal levels adjacent to pathologically involved nodal levels, based on the discretion of the treating oncologist
  Arms: Arm 2: SBRT arm
Radiation: Standard Radiation — Patients will receive daily conventional fractionation radiation over 4 or 6-6.5 weeks based on the treating oncologist's discretion. The below dose levels are recommended in the following clinical scenarios but may be modified per institutional standards: 20-fraction regimen or 30 to 33-fraction regimen
  Arms: Arm 1: Control

SUMMARY:
The purpose of this study is to compare the effectiveness and side effects of stereotactic radiotherapy (5 sessions) against conventional (standard) radiotherapy (20-30 sessions) for the treatment of skin cancer involving the head and neck after surgical resection.

Stereotactic radiotherapy works in the same way that conventional (standard) radiotherapy does to kill cancer cells by damaging their genetic material and stopping the cancer cells from making copies of themselves.

This study will help the study doctors find out if this different approach is the same, better, or worse than the standard of care for your cancer.

DETAILED DESCRIPTION:
This study is a phase II randomized trial where patients will be randomized in a 1:2 ratio to standard of care treatment with conventional fractionation PORT (Arm 1) vs. ultrahypofractionated stereotactic PORT (Arm 2). Patients will be stratified by pathologic nodal status (pN1 vs. pN2-pN3) per the American Joint Committee on Cancer (AJCC) 8th edition staging and use of immunotherapy (classified as neoadjuvant immunotherapy (with or without adjuvant immunotherapy) vs. planned for adjuvant immunotherapy only vs. no immunotherapy. Patients randomized to Arm 2 will be also compared to historical control data for primary endpoint of tumor local control at 2-years.

The objective of this study is to assess the clinical efficacy, toxicity and QOL of ultra-hypofractionated SABR compared to conventional fractionation for adjuvant radiation following resection of locally advanced, node-positive cutaneous SCC of the head and neck.

Primary endpoint

- Tumor control within the irradiated field at 2 years following adjuvant radiation completion defined as absence of clinical, radiographic or biopsy-proven recurrence within the irradiated field

Secondary endpoints

* Regional recurrence
* Disease-free survival (DFS)
* Overall survival (OS)
* Rate of salvage treatment (surgery in the ipsilateral neck) and freedom from unsalvageable recurrence in the ipsilateral parotid gland or neck
* Radiation-associated toxicity based on the Common Terminology Criteria for Adverse Events(CTCAE) version 5.0
* Patient-reported outcomes using the MD Anderson Symptom Inventory for Head and Neck Cancer (MDASI-HN) and the EuroQOL 5-Dimension 5-Level (EQ-5D-5L) questionnaires

ELIGIBILITY:
Inclusion criteria

* Age ≥ 18 years
* Patient able to provide informed consent
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Patient is a candidate for curative intent treatment
* Patient is able to comprehend English adequately to complete patient reported outcome questionnaires
* Biopsy-confirmed cutaneous SCC
* Definitive resection of a primary cutaneous tumor within the head and neck
* Tumor stage T1-T4 (AJCC 8th edition); or tumor stage unknown (T0/Tx) with a positive intraparotid, peri-parotid or cervical node that is assumed to be from a head and neck cutaneous SCC by the treating oncologist
* Nodal stage N1-N3 (AJCC 8th edition)
* At least 1 indication for adjuvant radiation, including:

  * T3 or T4 tumor stage
  * Lymphovascular invasion (LVI)
  * Perineural invasion (PNI)
  * Positive or close (≤ 3 mm) margin
  * ≥ 1 positive intraparotid, peri-parotid or cervical lymph node
  * Multiple local recurrences or multi-focal disease
* Neoadjuvant or adjuvant immunotherapy is allowed

Exclusion criteria

* Definite metastatic disease at diagnosis
* Pregnant or breastfeeding women
* Significant health conditions or contraindications to receiving surgery and radiation
* History of previous head and neck cancer within 5 years, except for localized skin cancers (i.e. no nodal or distant spread)
* Prior head and neck radiation involving the ipsilateral parotid or neck. However, prior radiation to the index skin cancer that has led to the parotid nodal disease being treated on this trial is allowed, as long as there is no overlap, or inconsequential overlap, in the judgement of the treating oncologist.
* Indications for contralateral neck radiation (i.e. contralateral or bilateral lymph nodes)
* Previous invasive malignancy within 5 years, unless controlled with no evidence of disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-10-21 (Actual); Primary Completion 2030-09-01 (Estimated); Study Completion 2035-09-01 (Estimated)

PRIMARY OUTCOMES:
Tumor control | 2 years
  Tumor control within the irradiated field at 2 years following adjuvant radiation completion defined as absence of clinical, radiographic or biopsy-proven recurrence within the irradiated field

SECONDARY OUTCOMES:
Regional recurrence | 2 years
  calculated as time from randomization to evidence of disease recurrence anywhere in the ipsilateral parotid gland or neck
Disease-free survival (DFS) | 2 years
  calculated as time from randomization to evidence of recurrence at any site, death from any cause, or last follow-up, whichever occurs first. New primary cutaneous SCC of the head or neck will not be counted towards DFS events.
Overall survival | 2 years
  calculated as time from randomization to death from any cause, or last follow-up, whichever occurs first.
Rate of salvage surgery | 2 years
  calculated as time from randomization to salvage surgery in the ipsilateral treated neck. Freedom from unsalvageable parotid/neck recurrence will be documented as time from randomization to evidence of recurrence in the ipsilateral parotid gland or neck that cannot be salvaged (either surgery or radiation), or last follow-up, whichever occurs first.
Radiation-associated toxicity | Baseline, during treatment, 2 weeks post treatment, 4 weeks post treatment, 3, 12, 18, 24 months post treatment, and yearly from years 2-5 after the end of radiation.
  Radiation-associated toxicity based on the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0, grade 2 or higher.
Patient-reported outcomes | Baseline, 3, 6, 12, 18, 24 months post-treatment and yearly from years 2-5 after the end of radiation.
  Patient-reported outcomes using the MD Anderson Symptom Inventory for Head and Neck Cancer (MDASI-HN) questionaries. The head and neck cancer specific symptoms are rated on a 0-10 scale to indicate the presence and severity of the symptoms. Lower scores represent better functioning and quality of life.
Patient Reported Outcome | Baseline, 3, 6, 12, 18, 24 months post-treatment and yearly from years 2-5 after the end of radiation.
  Patient reported outcome using the Euro QOL 5-Dimension 5-Level (EQ-5D-5L) questionnaire. EQ-5D-5L is a widely used questionnaire for measuring health-related quality of life, assessing five key health areas (Mobility, Self-care, Usual Activities, Pain/Discomfort, Anxiety/Depression) with five levels of severity (no to extreme problems) and a self-rated health scale (EQ-VAS) for overall well-being, helping evaluate treatments and health interventions.

CONTACTS AND LOCATIONS:
Locations (1):
- Verspeeten Family Cancer Centre, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Culbert M, Bidermann G, Wallace AS. Decisional preferences and satisfaction with short-course radiation for breast cancer. JCO. 2018;36(30_suppl):193-193. doi:10.1200/JCO.2018.36.30_suppl.193
- [Background] National Comprehensive Cancer Network Squamous Cell Skin Cancer (version 1.2024). https://www.nccn.org/professionals/physician_gls/pdf/squamous.pdf. Accessed 24 August 2024.
- [Background] National Cancer Institute-Common Toxicity Criteria Adverse Events Version 5. Published 2017. https://ctep.cancer.gov/protocolDevelopment/electronic_applications/docs/CTCAE_v5_Quick_Refer ence_8.5x11.pdf. Accessed 25 August 2024.
- [Background] Harris PA, Taylor R, Thielke R, Payne J, Gonzalez N, Conde JG. Research electronic data capture (REDCap)--a metadata-driven methodology and workflow process for providing translational research informatics support. J Biomed Inform. 2009 Apr;42(2):377-81. doi: 10.1016/j.jbi.2008.08.010. Epub 2008 Sep 30. PMID 18929686
- [Background] Hatswell A, Freemantle N, Baio G, Lesaffre E, van Rosmalen J. Summarising salient information on historical controls: A structured assessment of validity and comparability across studies. Clin Trials. 2020 Dec;17(6):607-616. doi: 10.1177/1740774520944855. Epub 2020 Sep 21. PMID 32957804
- [Background] Pocock SJ. The combination of randomized and historical controls in clinical trials. J Chronic Dis. 1976 Mar;29(3):175-88. doi: 10.1016/0021-9681(76)90044-8. No abstract available. PMID 770493
- [Background] Ringash J, O'Sullivan B, Bezjak A, Redelmeier DA. Interpreting clinically significant changes in patient-reported outcomes. Cancer. 2007 Jul 1;110(1):196-202. doi: 10.1002/cncr.22799. PMID 17546575
- [Background] Yao JJ, Zhou GQ, Jin YN, Zhang WJ, Lin L, Yu XL, Shao JY, Ma J, Sun Y. Predictors of Mastoiditis after Intensity-Modulated Radiotherapy in Nasopharyngeal Carcinoma: A Dose-Volume Analysis. J Cancer. 2016 Jan 8;7(3):276-82. doi: 10.7150/jca.13183. eCollection 2016. PMID 26918040
- [Background] Diao K, Nguyen TP, Moreno AC, Reddy JP, Garden AS, Wang CH, Tung S, Wang C, Wang XA, Rosenthal DI, Fuller CD, Gunn GB, Frank SJ, Morrison WH, Shah SJ, Lee A, Spiotto MT, Su SY, Ferrarotto R, Phan J. Stereotactic body ablative radiotherapy for reirradiation of small volume head and neck cancers is associated with prolonged survival: Large, single-institution, modern cohort study. Head Neck. 2021 Nov;43(11):3331-3344. doi: 10.1002/hed.26820. Epub 2021 Jul 16. PMID 34269492
- [Background] Grimm J, Vargo JA, Mavroidis P, Moiseenko V, Emami B, Jain S, Caudell JJ, Clump DA, Ling DC, Das S, Moros EG, Vinogradskiy Y, Xue J, Heron DE. Initial Data Pooling for Radiation Dose-Volume Tolerance for Carotid Artery Blowout and Other Bleeding Events in Hypofractionated Head and Neck Retreatments. Int J Radiat Oncol Biol Phys. 2021 May 1;110(1):147-159. doi: 10.1016/j.ijrobp.2020.12.037. Epub 2021 Feb 11. PMID 33583641
- [Background] Hanna GG, Murray L, Patel R, Jain S, Aitken KL, Franks KN, van As N, Tree A, Hatfield P, Harrow S, McDonald F, Ahmed M, Saran FH, Webster GJ, Khoo V, Landau D, Eaton DJ, Hawkins MA. UK Consensus on Normal Tissue Dose Constraints for Stereotactic Radiotherapy. Clin Oncol (R Coll Radiol). 2018 Jan;30(1):5-14. doi: 10.1016/j.clon.2017.09.007. Epub 2017 Oct 13. PMID 29033164
- [Background] Ng SP, Wang H, Pollard C 3rd, Nguyen T, Bahig H, Fuller CD, Gunn GB, Garden AS, Reddy JP, Morrison WH, Shah S, Rosenthal DI, Frank SJ, Guha-Thakurta N, Ferrarotto R, Hanna EY, Su SY, Phan J. Patient Outcomes after Reirradiation of Small Skull Base Tumors using Stereotactic Body Radiotherapy, Intensity Modulated Radiotherapy, or Proton Therapy. J Neurol Surg B Skull Base. 2020 Dec;81(6):638-644. doi: 10.1055/s-0039-1694052. Epub 2019 Jul 31. PMID 33381367
- [Background] Gerhard SG, Palma DA, Arifin AJ, Louie AV, Li GJ, Al-Shafa F, Cheung P, Rodrigues GB, Bassim CW, Corkum MT. Organ at Risk Dose Constraints in SABR: A Systematic Review of Active Clinical Trials. Pract Radiat Oncol. 2021 Jul-Aug;11(4):e355-e365. doi: 10.1016/j.prro.2021.03.005. PMID 34217495
- [Background] Nichols AC, Lang P, Prisman E, Berthelet E, Tran E, Hamilton S, Wu J, Fung K, de Almeida JR, Bayley A, Goldstein DP, Eskander A, Husain Z, Bahig H, Christopoulous A, Hier M, Sultanem K, Richardson K, Mlynarek A, Krishnan S, Le H, Yoo J, MacNeil SD, Mendez A, Winquist E, Read N, Venkatesan V, Kuruvilla S, Warner A, Mitchell S, Corsten M, Rajaraman M, Johnson-Obaseki S, Eapen L, Odell M, Chandarana S, Banerjee R, Dort J, Matthews TW, Hart R, Kerr P, Dowthwaite S, Gupta M, Zhang H, Wright J, Parker C, Wehrli B, Kwan K, Theurer J, Palma DA. Treatment de-escalation for HPV-associated oropharyngeal squamous cell carcinoma with radiotherapy vs. trans-oral surgery (ORATOR2): study protocol for a randomized phase II trial. BMC Cancer. 2020 Feb 14;20(1):125. doi: 10.1186/s12885-020-6607-z. PMID 32059705
- [Background] Nichols AC, Yoo J, Hammond JA, Fung K, Winquist E, Read N, Venkatesan V, MacNeil SD, Ernst DS, Kuruvilla S, Chen J, Corsten M, Odell M, Eapen L, Theurer J, Doyle PC, Wehrli B, Kwan K, Palma DA. Early-stage squamous cell carcinoma of the oropharynx: radiotherapy vs. trans-oral robotic surgery (ORATOR)--study protocol for a randomized phase II trial. BMC Cancer. 2013 Mar 20;13:133. doi: 10.1186/1471-2407-13-133. PMID 23514246
- [Background] Siu LL, Waldron JN, Chen BE, Winquist E, Wright JR, Nabid A, Hay JH, Ringash J, Liu G, Johnson A, Shenouda G, Chasen M, Pearce A, Butler JB, Breen S, Chen EX, FitzGerald TJ, Childs TJ, Montenegro A, O'Sullivan B, Parulekar WR. Effect of Standard Radiotherapy With Cisplatin vs Accelerated Radiotherapy With Panitumumab in Locoregionally Advanced Squamous Cell Head and Neck Carcinoma: A Randomized Clinical Trial. JAMA Oncol. 2017 Feb 1;3(2):220-226. doi: 10.1001/jamaoncol.2016.4510. PMID 27930762
- [Background] A Phase III Study of Postoperative Radiation Therapy (IMRT) +/- Cetuximab for Locally-Advanced Resected Head and Neck Cancer. Published online August 8, 2009. Accessed August 15, 2024. https://clinicaltrials.gov/study/NCT00956007
- [Background] Gillison ML, Trotti AM, Harris J, Eisbruch A, Harari PM, Adelstein DJ, Jordan RCK, Zhao W, Sturgis EM, Burtness B, Ridge JA, Ringash J, Galvin J, Yao M, Koyfman SA, Blakaj DM, Razaq MA, Colevas AD, Beitler JJ, Jones CU, Dunlap NE, Seaward SA, Spencer S, Galloway TJ, Phan J, Dignam JJ, Le QT. Radiotherapy plus cetuximab or cisplatin in human papillomavirus-positive oropharyngeal cancer (NRG Oncology RTOG 1016): a randomised, multicentre, non-inferiority trial. Lancet. 2019 Jan 5;393(10166):40-50. doi: 10.1016/S0140-6736(18)32779-X. Epub 2018 Nov 15. PMID 30449625
- [Background] Hu M, Kim ANH, Emeto TI, Collins M, Chopping A, Lin C. Metastatic cutaneous squamous cell carcinoma to the parotid: Adjuvant radiotherapy and treatment outcomes. J Med Radiat Sci. 2023 Jun;70(2):161-170. doi: 10.1002/jmrs.650. Epub 2023 Feb 15. PMID 36790039
- [Background] Hong TS, Kriesel KJ, Hartig GK, Harari PM. Parotid area lymph node metastases from cutaneous squamous cell carcinoma: implications for diagnosis, treatment, and prognosis. Head Neck. 2005 Oct;27(10):851-6. doi: 10.1002/hed.20256. PMID 16114004
- [Background] Coombs AC, Butler A, Allison R. Metastatic cutaneous squamous cell carcinoma of the parotid gland: prognostic factors. J Laryngol Otol. 2018 Mar;132(3):264-269. doi: 10.1017/S0022215117001323. Epub 2017 Jul 5. PMID 28677515
- [Background] Chen AM, Grekin RC, Garcia J, Bucci MK, Margolis LW. Radiation therapy for cutaneous squamous cell carcinoma involving the parotid area lymph nodes: dose and volume considerations. Int J Radiat Oncol Biol Phys. 2007 Dec 1;69(5):1377-80. doi: 10.1016/j.ijrobp.2007.05.005. Epub 2007 Aug 8. PMID 17689882
- [Background] Voruganti IS, Poon I, Husain ZA, Bayley A, Barnes EA, Zhang L, Chin L, Erler D, Higgins K, Enepekides D, Eskander A, Karam I. Stereotactic body radiotherapy for head and neck skin cancer. Radiother Oncol. 2021 Dec;165:1-7. doi: 10.1016/j.radonc.2021.10.004. Epub 2021 Oct 11. PMID 34648871
- [Background] Biau J, Thivat E, Millardet C, Saroul N, Pham-Dang N, Molnar I, Pereira B, Durando X, Bourhis J, Lapeyre M. A multicenter prospective phase II study of postoperative hypofractionated stereotactic body radiotherapy (SBRT) in the treatment of early-stage oropharyngeal and oral cavity cancers with high risk margins: the STEREO POSTOP GORTEC 2017-03 trial. BMC Cancer. 2020 Aug 5;20(1):730. doi: 10.1186/s12885-020-07231-3. PMID 32758188
- [Background] Mohamad I, Karam I, El-Sehemy A, Abu-Gheida I, Al-Ibraheem A, Al-Assaf H, Aldehaim M, Alghamdi M, Alotain I, Ashour M, Bushehri A, ElHaddad M, Hosni A. The Evolving Role of Stereotactic Body Radiation Therapy for Head and Neck Cancer: Where Do We Stand? Cancers (Basel). 2023 Oct 16;15(20):5010. doi: 10.3390/cancers15205010. PMID 37894377
- [Background] Murray Brunt A, Haviland JS, Wheatley DA, Sydenham MA, Alhasso A, Bloomfield DJ, Chan C, Churn M, Cleator S, Coles CE, Goodman A, Harnett A, Hopwood P, Kirby AM, Kirwan CC, Morris C, Nabi Z, Sawyer E, Somaiah N, Stones L, Syndikus I, Bliss JM, Yarnold JR; FAST-Forward Trial Management Group. Hypofractionated breast radiotherapy for 1 week versus 3 weeks (FAST-Forward): 5-year efficacy and late normal tissue effects results from a multicentre, non-inferiority, randomised, phase 3 trial. Lancet. 2020 May 23;395(10237):1613-1626. doi: 10.1016/S0140-6736(20)30932-6. Epub 2020 Apr 28. PMID 32580883
- [Background] Raldow AC, Chen AB, Russell M, Lee PP, Hong TS, Ryan DP, Cusack JC, Wo JY. Cost-effectiveness of Short-Course Radiation Therapy vs Long-Course Chemoradiation for Locally Advanced Rectal Cancer. JAMA Netw Open. 2019 Apr 5;2(4):e192249. doi: 10.1001/jamanetworkopen.2019.2249. PMID 30977859
- [Background] Newman JG, Hall MA, Kurley SJ, Cook RW, Farberg AS, Geiger JL, Koyfman SA. Adjuvant therapy for high-risk cutaneous squamous cell carcinoma: 10-year review. Head Neck. 2021 Sep;43(9):2822-2843. doi: 10.1002/hed.26767. Epub 2021 Jun 7. PMID 34096664
- [Background] Melo GM, Guilherme LH, Palumbo MDN, Rosano M, Neves MCD, Callegari FM, Abrahao M, Cervantes O. Parotidectomy and neck dissection in locally advanced and relapsed cutaneous squamous cell carcinoma of the head and neck region. Braz J Otorhinolaryngol. 2022 Nov-Dec;88 Suppl 4(Suppl 4):S152-S162. doi: 10.1016/j.bjorl.2021.11.007. Epub 2021 Dec 10. PMID 35042657
- [Background] Veness MJ, Palme CE, Smith M, Cakir B, Morgan GJ, Kalnins I. Cutaneous head and neck squamous cell carcinoma metastatic to cervical lymph nodes (nonparotid): a better outcome with surgery and adjuvant radiotherapy. Laryngoscope. 2003 Oct;113(10):1827-33. doi: 10.1097/00005537-200310000-00031. PMID 14520114
- [Background] O'Brien CJ, McNeil EB, McMahon JD, Pathak I, Lauer CS, Jackson MA. Significance of clinical stage, extent of surgery, and pathologic findings in metastatic cutaneous squamous carcinoma of the parotid gland. Head Neck. 2002 May;24(5):417-22. doi: 10.1002/hed.10063. PMID 12001070
- [Background] O'Brien CJ, McNeil EB, McMahon JD, Pathak I, Lauer CS. Incidence of cervical node involvement in metastatic cutaneous malignancy involving the parotid gland. Head Neck. 2001 Sep;23(9):744-8. doi: 10.1002/hed.1106. PMID 11505484
- [Background] Hinerman RW, Indelicato DJ, Amdur RJ, Morris CG, Werning JW, Vaysberg M, Kirwan J, Mendenhall WM. Cutaneous squamous cell carcinoma metastatic to parotid-area lymph nodes. Laryngoscope. 2008 Nov;118(11):1989-96. doi: 10.1097/MLG.0b013e318180642b. PMID 18849863
- [Background] Thom JJ, Moore EJ, Price DL, Kasperbauer JL, Starkman SJ, Olsen KD. The Role of Total Parotidectomy for Metastatic Cutaneous Squamous Cell Carcinoma and Malignant Melanoma. JAMA Otolaryngol Head Neck Surg. 2014 Jun;140(6):548-54. doi: 10.1001/jamaoto.2014.352. PMID 24722863
- [Background] Gregoire V, Ang K, Budach W, Grau C, Hamoir M, Langendijk JA, Lee A, Le QT, Maingon P, Nutting C, O'Sullivan B, Porceddu SV, Lengele B. Delineation of the neck node levels for head and neck tumors: a 2013 update. DAHANCA, EORTC, HKNPCSG, NCIC CTG, NCRI, RTOG, TROG consensus guidelines. Radiother Oncol. 2014 Jan;110(1):172-81. doi: 10.1016/j.radonc.2013.10.010. Epub 2013 Oct 31. PMID 24183870
- [Background] Bradley PJ. Parotid lymph nodes in primary malignant salivary neoplasms. Curr Opin Otolaryngol Head Neck Surg. 2022 Apr 1;30(2):99-106. doi: 10.1097/MOO.0000000000000772. PMID 35255046
- [Background] Likhacheva A, Awan M, Barker CA, Bhatnagar A, Bradfield L, Brady MS, Buzurovic I, Geiger JL, Parvathaneni U, Zaky S, Devlin PM. Definitive and Postoperative Radiation Therapy for Basal and Squamous Cell Cancers of the Skin: Executive Summary of an American Society for Radiation Oncology Clinical Practice Guideline. Pract Radiat Oncol. 2020 Jan-Feb;10(1):8-20. doi: 10.1016/j.prro.2019.10.014. Epub 2019 Dec 9. PMID 31831330
- [Background] Eggermont CJ, Eggermont AMM. Shifting landscape in skin cancer incidence: the rising tide of cutaneous squamous cell carcinoma and potential implications for prevention. Br J Dermatol. 2024 Mar 15;190(4):460-461. doi: 10.1093/bjd/ljad480. No abstract available. PMID 38099564